CLINICAL TRIAL: NCT04757246
Title: RESPECT Heart Failure- RESpiratory Pattern Evaluation in Clinical Trials for HF
Acronym: RESPECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding from Sponsor did not come through
Sponsor: WakeMed Health and Hospitals (Other)
Responsible Party: Principal Investigator, Stuart Russell, M.D., Principal Investigator, WakeMed Health and Hospitals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1705978
Record Dates: First submitted 2021-01-21; First posted 2021-02-17 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): Stable outpatients without implantable devices
  Interventions: Other: MouthLab Device
- Cohort 2 (Other): Stable outpatients with Boston Scientific pacemakers or defibrillators with Heart Logic capability
  Interventions: Other: MouthLab Device
- Cohort 3 (Other): Stable outpatients with implantable CardioMEMS devices
  Interventions: Other: MouthLab Device

INTERVENTIONS:
Other: MouthLab Device — Use of MouthLab system

SUMMARY:
The goal is to evaluate the trends in MouthLab parameters (respiration rate, temperature, pulse rate, electrocardiogram rhythm, blood pressure, oxygen saturation heart rate and basic lung function measures) in patients with decompensated heart failure and how these measurements change in response to decongestion. The research will test the ability of the MouthLab device to predict clinical decompensation in patients with known heart failure and to reduce the number of hospital readmissions based on the treatment guided by MouthLab device data.

DETAILED DESCRIPTION:
Heart failure (HF) is becoming increasingly recognized with an estimated worldwide prevalence of >37.7 million individuals. In the United States alone, there are over 5 million patients with HF which is expected to increase to over 8 million by 2030. Despite advances in medical therapies and technology, HF remains the leading cause of hospitalization among adults and the elderly. By 2030, the medical costs of HF are expected to rise from $20.9 billion to $53.1 billion, with nearly 80% of the projected increased expenses attributes to hospitalization costs. As such, it is imperative to develop new technologies and treatment options to impact the HF epidemic.

The majority of HF hospital admissions are due to volume overload. Stiffened and/or weakened myocardium predisposes patients to the accumulation of extracellular fluid resulting in increased intracardiac filling pressures and symptoms of congestion (edema, dyspnea and orthopnea). Accurate assessment of a patient's volume status remains clinically challenging at times. While there have been technological advances in the outpatient monitoring of volume status through thoracic impedance and pulmonary artery pressure monitoring, there are no validated, non-implantable options for monitoring volume status outside of the physical exam.

Aidar Health's MouthLab device is a non-invasive, hand-held, home monitoring tool that measures multiple medical parameters such as - Temperature, Blood Pressure, Heart Rate, Heart Rate Variability, Pulse Rate, SpO2, single-lead ECG, Respiratory Rate, Breathing Pattern/Respiratory Flow Cycle Morphology, and basic lung functions (FEV1, FVC, FEV1/FVC, PEF) in 30 seconds.

The investigators believe that the MouthLab device holds the potential to identify changes in volume status through measurements such as pulse rate, oxygen saturation, respiratory flow and lung function and accurately predict decompensation in patients with chronic HF. The investigators propose the following outline of clinical studies to evaluate the utility of the MouthLab device in HF.

ELIGIBILITY:
Inpatient Sub-Study Eligibility Criteria

Inclusion Criteria

1. Adults aged ≥ 18 years old
2. Willing and able to provide informed consent
3. Admitted within previous 24 hours with HF exacerbation requiring intravenous diuretic therapy (reduced or preserved ejection fraction)
4. English speaking

Exclusion Criteria

1. Currently on dialysis
2. Patients with acute coronary syndrome
3. Currently on hospice
4. Have a heart transplant or left ventricular assist device

   * Outpatient Sub-Study Eligibility Criteria

Inclusion Criteria

1. Adults aged ≥ 18 years old
2. Willing and able to provide informed consent
3. Patients presenting to the clinic and not being admitted to the hospital, who have been admitted for a HF exacerbation within the past 6 months, OR patients being discharged from a HF exacerbation related inpatient hospitalization
4. For inclusion in Cohort 2, patients must have Boston Scientific pacemaker or defibrillator with Heart Logic capability
5. For inclusion in Cohort 3, patients must have implantable CardioMEMS device
6. Patients currently on inotropes
7. English speaking

Exclusion Criteria

1. Currently on dialysis
2. Currently on hospice
3. Have a heart transplant or left ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Evaluate trends of respiration rate per minute | 6 months
  Respiration rate measured by breaths taken per minute
Aidar Questionnaire to Evaluate Patient Perception of Heart Failure | 6 months
  The Aidar Questionnaire will be used to determine patient perception of severity of heart failure.
Evaluate trends of temperature measured in Fahrenheit | 6 months
  Temperature
Evaluate trends of pulse rate per minute | 6 month
  Pulse rate
Evaluating the P wave of electrocardiogram in milliseconds | 6 months
  P wave on electrocardiogram will be measured to determine heart rhythm
Evaluating the QRS complex on electrocardiogram in milliseconds | 6 months
  QRS complex will be measured to determine heart rhythm
Evaluating the T wave on electrocardiogram in milliseconds | 6 months
  T wave will be measured to determine heart rhythm
Evaluate trends of blood pressure measured in mm/Hg | 6 months
  Blood pressure
Evaluate trends of blood oxygen saturation (SpO2) in percentage | 6 months
  blood oxygen saturation (SpO2)
Measuring FEV1 (Forced Expiratory Volume) in Liters | 6 months
  Determining Lung Function
Measuring FVC (Forced Vital Capacity) in Liters | 6 months
  Determining Lung Function
Measuring FEV1/FVC as a ratio | 6 months
  Determining Lung Function
Measuring PEF (Peak Expiratory Flow) in Liters/second | 6 months
  Determining Lung Function

CONTACTS AND LOCATIONS:
Locations (1):
- WakeMed Health and Hospitals, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Result] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Result] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Result] Felker GM, Ellison DH, Mullens W, Cox ZL, Testani JM. Diuretic Therapy for Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 17;75(10):1178-1195. doi: 10.1016/j.jacc.2019.12.059. PMID 32164892
- [Result] Guyatt GH, Nogradi S, Halcrow S, Singer J, Sullivan MJ, Fallen EL. Development and testing of a new measure of health status for clinical trials in heart failure. J Gen Intern Med. 1989 Mar-Apr;4(2):101-7. doi: 10.1007/BF02602348. PMID 2709167
- [Result] Garin O, Ferrer M, Pont A, Rue M, Kotzeva A, Wiklund I, Van Ganse E, Alonso J. Disease-specific health-related quality of life questionnaires for heart failure: a systematic review with meta-analyses. Qual Life Res. 2009 Feb;18(1):71-85. doi: 10.1007/s11136-008-9416-4. Epub 2008 Dec 4. PMID 19052916